CLINICAL TRIAL: NCT02266537
Title: A Parallel Group Study With Three Different α-antagonists and Placebo Once Daily Over Three Weeks to Assess Their Influence on the Extent of Weekly Phenylephrine-induced Mydriasis at Three Different Concentrations of Phenylephrine in Healthy Male Volunteers
Brief Title: Study to Assess the Influence of Three Different α-antagonists and Placebo on the Extent of Weekly Phenylephrine-induced Mydriasis at Three Different Concentrations of Phenylephrine in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 527.70
Record Dates: First submitted 2014-10-16; First posted 2014-10-17 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Tamsulosin; AlnA protein, Acinetobacter radioresistens; alfuzosin; Doxazosin

ARMS (4):
- Tamsulosin (Experimental)
  Interventions: Drug: Tamsulosin
- Alfuzosin (Experimental)
  Interventions: Drug: Alfuzosin
- Doxazosin (Experimental)
  Interventions: Drug: Doxazosin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamsulosin
  Other Names: Alna®
  Arms: Tamsulosin
Drug: Alfuzosin
  Other Names: Uroxatral® uno
  Arms: Alfuzosin
Drug: Doxazosin
  Other Names: Cardular PP Uro®
  Arms: Doxazosin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study was aimed to evaluate the pharmacological effect of different α-antagonists on phenylephrine induced pupil size in healthy male volunteers as pharmacological basis for Intraoperative floppy iris syndrome (IFIS)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* Age ≥ 21 and ≤ 55 years
* Body Mass Index (BMI) ≥ 18.5 and ≤ 29.9 kg/m2
* Signed and dated written informed consent in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and Electrocardiogram (ECG)) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24:00 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study or during the study
* Use of any drugs which might influence the results of the trial up to seven days prior to enrolment in the study or during the study
* Participation in another trial with an investigational drug (≤ two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on in-house trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (≥ 100 mL within four weeks prior to administration or during the trial)
* Any laboratory value outside the clinically accepted reference range
* Excessive physical activities within the last week before the trial or during the trial

The following exclusion criteria are of special interest for this study:

* Hypersensitivity to any alpha agonist, or to phenylephrine
* Supine blood pressure at screening of systolic < 110 mmHg and diastolic < 60 mmHg
* Ophthalmological criteria:

  * Corrected visual acuity < 0.5
  * Refractive Error with a spherical equivalent > +6 or smaller - 6 D
  * Elevated intraocular pressure (higher than 22 mmHg)
  * Relevant anisocoria or pupil deformation
  * History of eye surgery apart from laser trabeculoplasty less than three months previously or extraocular surgery such as strabismus surgery
  * Topical ocular medication influencing IOP (intraocular pressure) or pupil size within 3 months prior to study-start

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2005-11; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Sum of changes from baseline in the mean pupil diameters | Baseline, 60 and 80 min after administration of phenylephrine (PE)

SECONDARY OUTCOMES:
Change from baseline in mean diameter of both pupils | Baseline, 60 and 80 min after administration of phenylephrine (PE)
Change from baseline in mean diameter of both pupils | one week after cessation of drug
Concentration of the analyte in plasma | Up to 29 days after first administration of α-antagonists
Number of participants with clinically significant changes in vital signs | Up to 8 days after last pupillometry
Number of participants with abnormal changes in clinical laboratory parameters | Up to 8 days after last pupillometry
Number of participants with Adverse Events | Up to 8 days after last pupillometry
Assessement of global tolerability by investigator on a 4 point scale | 8 days after last pupillometry